CLINICAL TRIAL: NCT03575130
Title: Prospective Single-centre Randomized Observer-blind Placebo-controlled Parallel-group Phase IIa Clinical Trial to Investigate the Safety and Efficacy of Ripasudil 0.4% Eye Drops After Descemetorhexis in Patients With Moderate to Advanced Fuchs Endothelial Corneal Dystrophy (FECD)
Brief Title: Ripasudil 0.4% Eye Drops in Fuchs Endothelial Corneal Dystrophy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-002490-19
Record Dates: First submitted 2018-06-08; First posted 2018-07-02 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Fuchs' Endothelial Dystrophy; Fuchs Dystrophy; Corneal Endothelial Dystrophy; Corneal Endothelial Cell Loss; Cornea Guttata
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Dystrophy, Posterior Polymorphous, 1; Corneal Endothelial Cell Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glanatec (Experimental)
  Interventions: Drug: Ripasudil eye drops; Procedure: Descemetorhexis
- Placebo (Placebo Comparator)
  Interventions: Drug: Optive eye drops; Procedure: Descemetorhexis

INTERVENTIONS:
Drug: Ripasudil eye drops — Rho-kinase-Inhibitor (IMP)
  Arms: Glanatec
Drug: Optive eye drops — Artificial tears (placebo)
  Arms: Placebo
Procedure: Descemetorhexis — Corneal endothelial cells are removed prior to IMP administration by Descemetorhexis.

SUMMARY:
The cornea forms our "window to the world". Hence, its transparency is of utmost importance for vision. Corneal endothelium plays a central role in the maintenance of a transparent corneal stroma. It limits stromal fluid uptake from the anterior chamber of the eye through the formation of tight junctions. Simultaneously, fluid is actively transported from corneal stroma into the anterior chamber. This maintains the corneal stroma in a state of relative dehydration, thereby ensuring a constant distance of stromal collagen lamellae to each other, which in turn forms the basis for transparency of this tissue. If however corneal endothelial function is impaired, stromal swelling leads to corneal clouding and loss of vision.

Fuchs endothelial corneal dystrophy represents the most common form of corneal dystrophy. It occurs sporadically, however in some cases autosomal dominant inheritance has been described. This condition leads to progressive loss of corneal endothelium (typically around the age of 50-60 years), causing visual impairment due to swelling and opacification of corneal stroma.

Cell culture experiments have been able to show that chemical inhibitors of Rho-Kinase promote corneal endothelial cell proliferation and reduce apoptosis, while topical application in an animal model promoted corneal endothelial wound healing. This has prompted the notion of using topical Rho-kinase-inhibitor treatment to support endothelial cell regeneration in Fuchs endothelial corneal dystrophy.

Since September 2014, Rho-kinase-inhibitor eye drops (ripasudil) are clinically available in Japan for reduction of intraocular pressure in Glaucoma patients. Ripasudil eye drops therefore represent a strong candidate for safe and effective adjunctive treatment in patients with Fuchs corneal endothelial cell dystrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject
2. Understanding of study procedures and willingness to abide by all procedures during the course of the study.
3. Age range: 18-70 years
4. Diagnosis of moderate to advanced FECD with central guttae and clinical relevant corneal endothelial cell loss of <1,000 cells/mm2 and clinical indication of surgical intervention (descemetorhexis) with or without accompanying cataract operation
5. Reduced visual acuity, defined as BCVA <20/30
6. Woman of childbearing potential must be using a highly effective method of birth control.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of serious adverse reaction within the observation period of 3 months after descemetorhexis. | 3 Months

SECONDARY OUTCOMES:
rate of adverse event, adverse reaction, serious adverse event, serious adverse reaction and suspected unexpected serious adverse reaction | within the observation period of 6 months
effect of ripasudil on corneal endothelial cell density (ECD) | within the observation period of 6 months
effect of ripasudil on corneal thickness | within the observation period of 6 months
effect of on visual acuity (BCVA) | within the observation period of 6 months
effect of ripasudil on contrast sensitivity | within the observation period of 6 months
assess the need of rescue therapy (DMEK) | within the observation period of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, University of Erlangen-Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No